CLINICAL TRIAL: NCT03500406
Title: Penile Lengthening Pre-Penile Prosthesis Implantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed subspecialties and no longer had access to main study population
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Landon W. Trost, Consultant, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-011052
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 - Control (Sham Comparator): No treatment will be administered and men will not have to delay their IPP procedure
  Interventions: Other: Control
- Group 2 - PTT 3x daily x 3 months (Experimental): Men will utilize penile traction therapy for 30 minutes three times daily for the 3 months prior to placement of their IPP
  Interventions: Device: RestoreX

INTERVENTIONS:
Device: RestoreX — Penile traction therapy in the straight position
  Arms: Group 2 - PTT 3x daily x 3 months
Other: Control — No treatment
  Arms: Group 1 - Control

SUMMARY:
This study is intended to utilize a novel, class I (ie. lowest risk, clinical studies not required) medical device to determine whether penile length can be increased in men prior to undergoing a penile prosthesis implantation procedure.

DETAILED DESCRIPTION:
Men with erectile dysfunction, unresponsive to conservative therapies, are recommended to undergo placement of an inflatable penile prosthesis (IPP); however, it is a common complaint post-operatively that their penis length is shorter than what it was previously.

Several attempts have been made by investigators to optimize penile length prior to placement of the penile prosthesis. Compared to other options, penile traction therapy (PTT) offers several potential advantages in that it is minimally-invasive, does not increase the morbidity of surgery, and has not been shown to result in any long-term side effects.

A new penile traction device (RestoreX® ) was created and funded through Mayo Ventures. Given the clinical issue of dissatisfaction with penile length post IPP, the potential role for PTT, and limited amount of data available, we sought to perform a clinical trial evaluating the effect of PTT on increasing the total length of prosthesis which can be inserted. We additionally sought to determine if PTT resulted in improved post-operative satisfaction on total penile length achieved.

To accomplish the study, a population of men from Mayo Clinic planning to undergo placement of an IPP will be enrolled and given the option to either join the control (no treatment) group or PTT group for 3 months prior to their procedure. Outcomes will be assessed prior to surgery and 3, 6, and 12 months post-procedure. Results are to be used with the intent to publish in a scientific journal.

ELIGIBILITY:
Inclusion Criteria

* Men undergoing placement of a penile prosthesis
* Must be the first time a penile prosthesis is implanted
* Undergoing implantation of a 3-piece inflatable penile prosthesis

Exclusion Criteria

* Prior ischemic priapism
* Any prior penile prosthesis surgeries
* Any prior penile surgeries other than circumcision
* Undergoing malleable penile prosthesis or Ambicor device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Landon W Trost, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Started | 4 | 20
Completed | 4 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months | Total
Number analyzed (Participants) | 4 | 20 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.9) | 63.1 (9.1) | 63.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 20 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 20 | 24

OUTCOME MEASURES:

1. Primary Outcome: Length Assessment of Penile Prosthesis Implanted
Description: The primary objective is to assess the length of the penile prosthesis inserted into subjects following completion of RestoreX® traction therapy compared to the control group (no treatment)
Time Frame: From baseline to 3 months
Population: Study was terminated due to PI change of subspecialties and no longer able to access the main study population. Sincere efforts were made but we were unable to collect data.
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Participant Compliance
Description: Compare Participant compliance with traction device
Time Frame: From baseline to 3 months
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Participant Satisfaction With Traction
Description: Compare patient reported satisfaction with use of traction device
Time Frame: From baseline to 3 months
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Events With Use of Traction
Description: Evaluate any adverse events with use of RestoreX® for penile lengthening.
Time Frame: From baseline to 3 months
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Operative Complications
Description: Compare intra- and/or post-operative complication rates.
Time Frame: 3, 6, 12 months post-operative
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Stretched Penile Length
Description: Compare pre- and post-operative stretched penile lengths
Time Frame: From baseline to 12 months
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Participant Satisfaction Penile Length
Description: Compare participant satisfaction scores including satisfaction with overall penile length
Time Frame: Baseline to 12 months post-operative
Population: as for outcome 1
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected three months post prosthesis implantation. However, this study was terminated due to PI change of subspecialties and no longer able to access the main study population. Sincere efforts were made but we were unable to collect data.
Arm/Group | Group 1 - Control | Group 2 - PTT 3x Daily x 3 Months
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/20
Other Adverse Events (participants affected / at risk) | 0/4 | 0/20

LIMITATIONS AND CAVEATS:
Study was terminated due to PI change of subspecialties and no longer able to access the main study population. Sincere efforts were made but we were unable to collect data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03500406/Prot_SAP_002.pdf